CLINICAL TRIAL: NCT06896929
Title: Comparison of Topical Permethrin 1 Day Verses 2 Day Application Versus Oral Ivermectin for Treatment of Scabies in Children Greater Than 6 Yrs of Age
Brief Title: Comparison of Permethrin and Ivermectin in Children Greater Than 6 Yrs Age for Treatment of Scabies
Acronym: not existed
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Children Hospital and Institute of Child Health, Lahore (Other)
Responsible Party: Principal Investigator, Sadaf Wazir, DR SADAF WAZIR, Children Hospital and Institute of Child Health, Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 715-24-10-2023ApprovedbyCHUCHS
Record Dates: First submitted 2025-03-20; First posted 2025-03-26 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2024-10

CONDITIONS: Scabies
Keywords: Comparison of permethrin and ivermectin in scabies
MeSH Terms: conditions — Scabies | interventions — Ivermectin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A (Experimental): Group A will be given Permethrin
  Interventions: Drug: Permethrin Cream, 5%
- Group B (Experimental): Group B will be given Permethrin 5% cream twice application
  Interventions: Drug: Permethrin Cream, 5%
- Group C (Experimental): Group C will be given Tab Ivermectin
  Interventions: Drug: Ivermectin 200 µg/kg

INTERVENTIONS:
Drug: Permethrin Cream, 5% — Permethrin 5% cream will be given as a single application
  Arms: Group A
Drug: Permethrin Cream, 5% — Permethrin Cream will be given as twice application
  Arms: Group B
Drug: Ivermectin 200 µg/kg — Group C will be given Tab Ivermectin
  Arms: Group C

SUMMARY:
Scabies is highly contagious,pruritic infestation of skin.Various treatment modalities have been used but search for ideal scabicide is ongoing.we wnt to coduct this study to compare the outcome of permethrin verses ivermectin in children for treatment of scabies .This randomized clinical trial will be done in children hospital lahore for 12 months.Sample size of 90 cases;30 in each group will be included through non probability consecutive sampling.Then patient will be randomly divided into 3 groups.In group A patient will be given 5% permethrin topical application to whole body single application. In Group B ,patients will be given topical permethrin for twice application 24 hrs appart ,In group C patients will be given Tablet Ivermectin single dose 200microgram/kg.Then patients will be examined after 2 weeks and 4 weeks for no of lesions and pruritis and cure will be labeled.All this information will be recorded on performa .Data will be entered and analysed by using SPSS version 26.Three groups will be compared for cure by using chi-square test.P value less than and equal to 0.05 will be considered as significant.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-15
* Both genders
* Diagnosed with scabies (as per operational definition)

Exclusion Criteria:

* Children with recurrent scabies on medical record
* Known allergy to ivermectin or permethrin.
* Widespread eczema or impetigo.
* Liver dysfunction or renal failure

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Cure of scabies. | 12 months
  Cure will be labeled if greater han 50% reduction in no of lesions and pruritis observed after 4 weeks of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Children Hospital Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/21860157/
- Available data/document: Clinical Study Report: permethrin — https://pubmed.ncbi.nlm.nih.gov/21860157/ — Comparison of permethrin and ivermectin in scabies was done